CLINICAL TRIAL: NCT06146361
Title: Vale+ Tu Salud: Corner-Based Randomized Trial to Test a Latino Day Laborer Program Adapted to Prevent COVID-19.
Brief Title: Vale+Tú Salud: Corner-Based Randomized Trial to Test a Latino Day Laborer Program Adapted to Prevent COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Maria Eugenia Fernandez-Esquer, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-20-1389 (phase 2); 1R01MD016328-01 (NIH)
Record Dates: First submitted 2023-11-22; First posted 2023-11-24 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
Keywords: Latino Day Laborers
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Cluster Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVID-19 Group Problem Solving (Experimental)
  Interventions: Behavioral: COVID-19 Group Problem Solving; Behavioral: Standard of Care
- Standard of Care (Active Comparator)
  Interventions: Behavioral: Standard of Care
- Group Problem Solving Plus Booster Session (Experimental)
  Interventions: Behavioral: COVID-19 Group Problem Solving; Behavioral: Standard of Care; Behavioral: Booster session

INTERVENTIONS:
Behavioral: COVID-19 Group Problem Solving — This group will have three core components to be delivered at the corner by trained data collectors. Interactive dialogue component that incorporates popular education activities aimed at developing social cohesion among LDLs, building awareness about COVID-19 risks and protective behaviors and developing a plan of action to reduce their and their peers' risk for COVID-19 transmission. Navigation Component will consist of providing information and linking LDLs with social service providers that can help buffer some of the social and economic effects of the COVID-19 pandemic and the "Multiplicador de salud"/Health Multiplier component that builds from the theoretical and practice-based method of mobilizing social networks and social support, defined as encouraging social networks to provide informational, emotional, appraisal, and instrumental support as cited in the Taxonomy of Behavior Change Methods.
  Arms: COVID-19 Group Problem Solving; Group Problem Solving Plus Booster Session
Behavioral: Standard of Care — This group will receive a COVID-19 prevention flyer and social resources list only
Behavioral: Booster session — Participants will have a 10 - 15 minute "booster' session about a week after engaging in the small group intervention. They will be contacted by phone and the booster will consist of brief prompts to engage participants in a discussion to encourage them to act on their personal commitments to protect themselves and others against COVID. They will also be encouraged to seek COVID related resources based on the information provided during the small group intervention.
  Arms: Group Problem Solving Plus Booster Session

SUMMARY:
The purpose of this study is to assess the extent to which LDL report increased adherence with COVID 19 mitigation practices 1 month post intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic or Latino
* Be present at the corner for the purposes of looking for work

Exclusion Criteria:

* Have not been previously hired to work at a corner
* Symptoms of COVID-19 in the previous 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 359 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Fernandez-Esquer, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: street corners
Groups:
- Group Problem Solving Plus Booster Session: COVID-19 Group Problem Solving: This group will have three core components to be delivered at the corner by trained data collectors. Interactive dialogue component that incorporates popular education activities aimed at developing social cohesion among LDLs, building awareness about COVID-19 risks and protective behaviors and developing a plan of action to reduce their and their peers' risk for COVID-19 transmission. Navigation Component will consist of providing information and linking LDLs with social service providers that can help buffer some of the social and economic effects of the COVID-19 pandemic and the "Multiplicador de salud"/Health Multiplier component that builds from the theoretical and practice-based method of mobilizing social networks and social support, defined as encouraging social networks to provide informational, emotional, appraisal, and instrumental support as cited in the Taxonomy of Behavior Change Methods.
  Standard of Care: This group will receive a COVID-19 prevention flyer and social resources list only
  Booster session: Participants will have a 10 - 15 minute "booster' session about a week after engaging in the small group intervention.
Period: Overall Study
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Started | 120; 8 street corners | 120; 8 street corners | 119; 8 street corners
Completed | 104; 8 street corners | 100; 8 street corners | 95; 8 street corners
Not Completed | 16; 0 street corners | 20; 0 street corners | 24; 0 street corners

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care | Total
Number analyzed (Participants) | 120 | 120 | 119 | 359
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: For age, data were not collected for 2 in the Group Problem Solving arm, for 2 in the Group Problem Solving Plus Booster Session arm, and for 2 in the Standard of Care arm.
  years
    number analyzed (Participants) | 118 | 118 | 117 | 353
    (all) | 43.4 (13.4) | 43.7 (12.4) | 40.3 (14.3) | 42.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 120 | 120 | 119 | 359
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 120 | 120 | 119 | 359
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120 | 120 | 119 | 359

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Compliant With COVID Vaccination Guidelines as Assessed by a Survey
Description: Measure of compliance with COVID vaccination guidelines.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Number analyzed (Participants) | 120 | 120 | 119
Participants | 30 | 28 | 33

2. Primary Outcome: Number of Participants Compliant With COVID Vaccination Guidelines as Assessed by a Survey
Description: Post test measure of compliance with COVID vaccination guidelines.
Time Frame: 4 weeks post intervention
Population: Data were not collected for 16 in the Group Problem Solving arm, for 20 in the Group Problem Solving plus Booster Session arm, and 24 in the Standard of Care arm--this is because these participants were lost to follow up at the 4-week timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Number analyzed (Participants) | 104 | 100 | 95
Participants | 59 | 53 | 53

3. Primary Outcome: Mask Wearing Frequency as Assessed by a Survey
Description: Mask Wearing frequency is reported as a score, ranging from 1-4, with a higher score indicating greater mask wearing frequency.
Time Frame: Baseline
Population: Data for this outcome measure were not collected for 2 in the Group Problem Solving arm and for 4 in the Group Problem Solving plus Booster Session arm--this is because these participants did not complete this survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Number analyzed (Participants) | 118 | 116 | 119
score on a scale | 2.050 (0.915) | 2.109 (0.836) | 1.927 (0.842)

4. Primary Outcome: Mask Wearing Frequency as Assessed by a Survey
Description: as for outcome 3
Time Frame: 4 weeks post intervention
Population: Data for this outcome measure were not collected for 16 in the Group Problem Solving arm, for 20 in the Group Problem Solving plus Booster Session arm, and for 24 in the Standard of Care arm--this is because these participants were lost to follow up at the 4-week timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Number analyzed (Participants) | 104 | 100 | 95
score on a scale | 1.720 (0.621) | 1.798 (0.567) | 1.632 (0.673)

5. Primary Outcome: Percentage of Participants Who Contacted an Agency About the Gold Card
Description: Percentage of participants who reported contacting a local community or health agency to request the Gold Card a local medical insurance for low income individuals living in Harris County.
Time Frame: 4 weeks post intervention
Population: For this outcome measure, data were collected only for those who called a number on the resource sheet--for the Group Problem Solving arm, 20 called a number; for the Group Problem Solving plus Booster Session arm, 22 called a number; and for the Standard of Care arm, 7 called a number.
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Number analyzed (Participants) | 20 | 22 | 7
Participants | 6 | 10 | 4

6. Primary Outcome: Percentage of Participants Who Reported Contacting the Agency for Assistance to Get Food
Description: Percentage of participants who reported seeking food assistance from a local community organization.
Time Frame: 4 weeks post intervention
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Number analyzed (Participants) | 20 | 22 | 7
Participants | 10 | 13 | 3

7. Primary Outcome: Percentage of Participants Who Reported Contacting the Agency for Assistance With Health Care Resources
Description: Percentage of participants who reported seeking medical assistance or health advice from a local clinic or community organization.
Time Frame: 4 weeks post intervention
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
Number analyzed (Participants) | 20 | 22 | 7
Participants | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: up to 30 days
Arm/Group | COVID-19 Group Problem Solving | Group Problem Solving Plus Booster Session | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 0/119
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 0/119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT06146361/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT06146361/ICF_001.pdf